CLINICAL TRIAL: NCT06708104
Title: Examining the Feasibility of an Outdoor Therapeutic Horse Carriage As a Perturbation -based Balance Training.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, Amir Haim, Principal investigator, Loewenstein Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOE-0010-24
Record Dates: First submitted 2024-11-18; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Balance Impairment; Accidental Fall
Keywords: Reactive balance; Perturbation training; Animal-assisted therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Outdoor horse-assisted perturbation training (Experimental): Outdoor perturbation training during Equine Dynamic Balance
  Interventions: Device: Outdoor horse-assisted perturbation training

INTERVENTIONS:
Device: Outdoor horse-assisted perturbation training — This is balance training in which a special carriage, i.e. a dynamic standing platform, is pulled by a horse on the outside surface, providing the trainee with multi-directional 3D balance perturbations that depend on the topography of the training area (various slopes and surface types), the horse walking speed, and its ability to stop, accelerate, and turns.

SUMMARY:
The proposed study is a prospective experimental single-arm pre-post study aiming to assess the effectiveness and feasibility of an outdoor therapeutic horse carriage, i.e., the Equine Dynamic Balance (EDB), as a form of reactive balance training. First, the investigators will describe the mechanical parameters of perturbations generated by the EDB's standing platform, including displacement, velocity and acceleration. Second, the investigators will assess the effect of EDB training on balance. Independent healthy young adults who do not suffer from balance impairments willing to participate in the study will be tested before and after EDB training, that will be delivered by standing on a dynamic therapeutic horse carriage pulled by a horse, to explore whether there are differences in balance control and balance reactions as a result of a 2-week EDB intervention program.

DETAILED DESCRIPTION:
Falls and fall-related injuries are serious and costly health problems, resulting in decreasing in quality of life, reducing mobility and independence and increasing morbidity and mortality. Most falls arise from events originating in the external environment when balance is lost unexpectedly due to a disruption to the base of support (BoS) directly (e.g., slips, trips during waking) or because of a rapid change in the center of mass (CoM) over the BoS (e.g., turns, being pushed). These situations are called externally induced balance perturbations. Reactively stepping and grasping something stable are effective strategies to increase the BoS, as they quickly decelerate the CoM motion, restoring equilibrium and averting falls.

Reactive balance is a critical basis for independent daily functioning; thus, it is a major training component in fall prevention programs. Reactive Balance Training (RBT) exposes participants to repeated unannounced external-induced balance perturbations in a safe and controlled environment aiming to specifically trigger, train and improve balance recovery skills. It was previously shown that adaptation to repeated-perturbation exposure can occur rapidly, even during a single-training session, suggesting that skill acquisition of reactive balance responses was accrued in a short amount of time.

RBT uses different stationary mechatronic systems that usually provide mediolateral or anteroposterior external perturbations during standing and treadmill walking. To date, RBTs lack a vertical component of balance disturbances additionally to a single type of perturbation direction may result in the limited real-life generalization.

the investigators were inspired by the growing body of research intervening humans with animal-assisted therapy, such as horses, to help people as they recover from physical and mental health conditions. Recent reviews of this novel therapeutic intervention indicate that participating in animal-assisted therapy has many benefits in motor and physical ability and also in mental and behavioral health among older, young and hospitalized patients. Therapeutic horseback riding (hippotherapy) intervention programs have been shown to improve balance, gait, and gross motor function in people with stroke, multiple sclerosis, children with cerebral palsy, as well as in older adults. However, traditional therapeutic horseback riding primarily occurs in a sitting position, which may not directly address balance training for situations in which balance losses occur in everyday lives (i.e., walking and standing). Therefore, introducing a dynamic horse-assisted balance training program in a standing position represents an innovative approach with added value.

To enhance the transfer of balance abilities from laboratory settings to real-world scenarios, the investigators propose a novel RBT program, The Equine Dynamic Balance (EDB). This program will introduce 3-dimensinal perturbations in various combined directions, targeting the change in BoS strategies through stepping and grasping as well as fixed-BoS strategies where feet remain stationary. The EDB is an outdoor therapeutic horse carriage, developed by "UDI Challenging Riding". This innovative apparatus serves as a platform for horse-assisted therapy for dynamic balance training while standing.

the investigators hypothesize that the Equine Dynamic Balance training could effectively integrate the principals of RBT with the health advantages of horse-assisted therapy, thereby establishing a novel effective form of RBT that provides multidirectional three-dimensional (3D) perturbations in a dynamic outdoor setting. This unique setting also enables elicitation of proprioception, vestibular, and visual stimuli in a similar way occurs during everyday balance disturbances. As far as the investigators know, this is the first outdoor animal-assisted RBT program, marking a proof-of-concept feasibility study.

Objectives: The overarching aim is to develop an EDB training program as a form of Reactive Balance Training and evaluate its feasibility in fostering the acquisition of reactive balance responses. The specific aims are as follows: 1) Describe the mechanical parameters of perturbations generated by the EDB's standing platform, including displacement, velocity and acceleration, under two conditions: a) Continuous riding, b) Fixed controlled spots of deceleration, stop, acceleration and turns along the horse track. 2) Assess the effect of EDB training on well-established biomechanical parameters of balance, i.e., stepping, and grasping responses, as well as step length and CoM path displacement, over a 2-week intervention program among healthy young adults.

Methods: This is a proof-of-concept feasibility study. Firstly, the investigators will characterize the 3D mechanical parameters of perturbations generated by the EDB's standing platform, including displacement, velocity and acceleration along the horse walking trail, and will describe the balance reactions following these perturbations. Secondly, the investigators will conduct a pre-post study to investigate the effects of a two-week EDB intervention program, including four sessions of 20-minute therapeutic horse carriage exercise, on reactive balance among healthy young adults. The study was approved by the Helsinki committee of Loewenstein Rehabilitation Hospital, Ra'anana, Israel (0010-24-LOE). All subjects will sign an informed consent statement.

Training program: the investigators will conduct four 20-minute EDB training sessions, consisting of 8 potential training levels, that gradually increase in difficulty based on balance and motor learning principles. This balance training is based on pulling the carriage on the outside surface, with its various slopes, that provides the trainee with multi-directional 3D balance perturbations that depend on the topography of the training area, the horse walking speed, and its ability to stop, accelerate, and turns. Therefore, this is a 3D balance perturbation training which includes various combinations of mediolateral, anterior-posterior, and vertical and rotatory perturbations in an outdoor dynamic environment.

Participants will stand on marked changeable footprints, in comfortable or wider standing positions, with feet at shoulder width or wider, respectively, on a dynamic platform of the carriage. They will be instructed to keep their balance and minimize their stepping and grasping responses while being exposed to a variety of balance perturbations, delivered by standing on a therapeutic horse carriage pulled by a horse. The horse will pull the carriage by walking in a figure of eight marked on the grass, consisting continuous riding parts and fixed sections of deceleration, stop, acceleration and turns for horse path and perturbations repeatability. Before the first training session and immediately after the end of the last fourth session pre- and post-test assessment will be performed.

Assessments: the investigators will measure and describe, pre-and post-tests and also during all 8 training levels, the mechanical parameters generated by the EDB's standing platform, and the following participants' balance reactions under two conditions: 1) continuous riding (i.e., spontaneous perturbations along the horse track); and 2) fixed spots of deceleration, stop, acceleration and turns (i.e., controlled perturbations).

the investigators will utilize two GoPro cameras and several inertial measurement units. The mechanical parameters will include 3D displacement, velocity and acceleration of the EDB's standing platform along the horse walking trail. The appropriate balance response to each perturbation will be measured observationally and quantitively by number of steps and grasping responses, and by total step path length and time of grasping the handrail, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young participants
* Adults aged 18-45 years
* Measuring between150-190 cm in stature, with a mass of less than 100 kg
* No neurological or vestibular or orthopedic mobility impairing conditions, and with no current musculoskeletal injury.

Exclusion Criteria:

* blindness or serious vestibular impairments (Meniere's disease, dizziness)
* an inability to ambulate independently
* symptomatic severe cardiovascular disease
* neurological disorders such as stroke, Parkinson's, or Multiple sclerosis
* orthopedic acute disorders requiring total hip or knee replacement
* severe rheumatoid arthritis; and/or (g) cancer (metastatic or under active treatment).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Reactive stepping response | change from baseline assessment (pre-test) to end of training program at 2 weeks (post-test).
  the total step path length is the sum of the total distance each foot travelled during perturbation until completing the recovery stepping response. It will be measured in centimeters.
Reactive stepping response during a training session | during a training session, an average of 20 minutes.
  the total step path length is the sum of the total distance each foot travelled during a perturbation until completing the recovery stepping response. It will be measured in centimetres.
The three-dimensional perturbation displacement | during a training session, an average of 20 minutes.
  The three-dimensional displacement, in three axes, of the dynamic platform in a balance perturbation. It will be measured in centimetres.
The three-dimensional perturbation velocity | during a training session, an average of 20 minutes.
  The three-dimensional velocity, in three axes, of the dynamic platform in a balance perturbation. It will be measured in meter per second (meter/second).
The three-dimensional perturbation acceleration | during a training session, an average of 20 minutes.
  The three-dimensional acceleration, in three axes, of the dynamic platform in a balance perturbation. It will be measured in meter/secound2.

SECONDARY OUTCOMES:
reactive grasping response | change from baseline assessment (pre-test) to end of training program at 2 weeks (post-test).
  : the total time a participant holds onto the safety handrail for recovering balance by grasping response. It will be measured in percentage, the fraction of the grasping time out of the total round time.
reactive grasping response during a training session | during a training session, an average of 20 minutes.
  the total time a participant holds onto the safety handrail for recovering balance by grasping response. It will be measured in percentage, the fraction of the grasping time out of the total round time.
total recovery time during a training session | during a training session, an average of 20 minutes.
  the time from perturbation onset to the end of balance recovery will be measured in milliseconds.
total recovery time | : change from baseline assessment (pre-test) to end of training program at 2 weeks (post-test).
  the time from perturbation onset to the end of balance recovery will be measured in milliseconds.

OTHER OUTCOMES:
satisfaction and subjective effects on balance in daily lives | at post-test, end of the 2-week training program.
  a 5-point-Likert-scale questionnaire (5=strongly agree): who much the exercise changes their balance in household and outdoor activities, exercise safety, challenging and diverse, customized to their ability, enjoyment, and whether they are interested in continuing the training program.

IPD SHARING:
Plan to Share IPD: No